CLINICAL TRIAL: NCT05599490
Title: BETTER Aging Trial: Brain Enhancement Training Towards Elders Resilience to Aging, Phase IIB
Brief Title: Brain Enhancement Training Towards Elders Resilience to Aging, Phase IIB
Acronym: BETTER Aging
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: University of Iowa (Other); The University of Texas at Dallas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSC-1024-22
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Age-related Cognitive Decline

STUDY DESIGN:
Masking Description: The Investigators and Assessors will be blinded to the previous treatment assignment of participants from the Phase II study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Treatment (Experimental): Computerized plasticity-based adaptive cognitive training requiring a total maximum of 50 treatment sessions, up to 5 sessions per week, 42 minutes per session.
  Interventions: Other: Computerized Plasticity-Based Adaptive Cognitive Training

INTERVENTIONS:
Other: Computerized Plasticity-Based Adaptive Cognitive Training — Forty-two minutes of training on computerized exercises that targets processing speed, memory and attention.
  Other Names: PACR-CT

SUMMARY:
This study aims to examine the longer-term benefits of a novel, neuroplasticity-based, computerized and web-deliverable training program (PACR-CT) five years from the initial 10 weeks of training from our Phase II study - Protocol #: PSC-0605-17 (Aim 1) and test the interactive effect of previous training and 10 weeks of booster training (Aim 2). Both the study and the software being investigated meet the criteria of Non-Significant Risk.

DETAILED DESCRIPTION:
This study will employ a single arm, open label design with use of the PACR-CT with all participants who completed the Phase II study, as well as approximately 60 new participants (with a goal of 40 completers) who are age-matched and untrained older adults. After consent, only the new, untrained participants will complete the screening visit. Then all participants will perform the pre-training visit (cognitive and functional assessments, MRI/fMRI and blood draw), followed by 10 weeks of training, and then followed by post-training visit (cognitive and functional assessments and MRI/fMRI).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 70 years of age or older
* Participant must be a fluent English speaker
* Participant must have adequate sensorimotor capacity to perform the program, including visual capacity adequate to read from a computer screen at a normal viewing distance, auditory capacity adequate to understand normal speech, and motor capacity adequate to control a computer mouse
* Participant must not have evidence of dementia as indicated by the Montreal Cognitive Assessment (MoCA)

Exclusion Criteria:

* Participant with any medical illnesses, injuries or conditions predisposing to imminent functional and/or cognitive decline
* Participant requiring caregiver assistance in dressing/personal hygiene
* Participant with severe visual deficits (including visual neglect, partial field cuts, anopias) and/or severe hearing deficit that would prevent use of the computerized treatment program
* Participant with recent participation of computer-delivered cognitive training within 2 years of consent
* Participant with claustrophobia or any other contraindication to MRI scanning
* Participant with inability to complete a 1-hour MRI
* Pregnant women
* Participant with any implanted devices above the waist (e.g., cardiac pacemaker or auto-defibrillators, neural pacemaker, aneurysm clips, cochlear implant, metallic bodies in the eye or central nervous system, any form of wires or metal devices that may concentrate radio frequency fields)
* Participants with active suicidal ideation with specific plan and intent or suicide-related behaviors within 2 months of consent as measured by the Columbia-Suicide Severity Rating Scale (C-SSRS)

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in performance on global cognitive composite score | At 5 years and at 3 months
  Change in performance on global cognitive composite score based on the average of all normalized assessment measures.

SECONDARY OUTCOMES:
Change in performance on processing speed composite score | At 5 years and at 3 months
  Change in performance on processing speed will be measured using the composite score created by averaging the z-scores of Pattern Comparison, Letter Comparison, and Digit Symbol Coding tasks.
Change in performance on working memory | At 5 years and at 3 months
  Change in performance on working memory will be measured using the composite score created by averaging the z-scores of Visual Short Term Memory and N-Back Tasks.
Changes in performance on episodic memory | At 5 years and at 3 months
  Change in performance on episodic memory will be measured using the composite score created by averaging the z-scores of Selective Reminding Task and Face Name Task.
Change in performance on executive function | At 5 years and at 3 months
  Change in performance on executive function will be measured using the composite score created by averaging the z-scores of Flanker Task and Task Switch (fMRI task).
Change in brain function | At 5 years and at 3 months
  Change in resting state functional connectivity will be measured by resting State T2*weighted EPI-BOLD, a 10-minute task-free BOLD contrast sequence consisting of 300 volumes (TR=2000 ms/TE=30ms) at 3.4mm3 in-plane resolution and 3mm slice thickness. Participants will be instructed to keep their eyes open and maintain attention on a central gray fixation cross on a black screen.
Change in brain structure | At 5 years and at 3 months
  3D T1-Weighted multi-echo MPRAGE. Morphometric analyses will be based on this MRI sequence (not accelerated because the reliability of acceleration for multi-site studies has not yet been established). We will achieve spatial resolution of 1 x 1 x 1 mm voxels.
Change in task-related brain activation | At 5 years and at 3 months
  Change in functional connectivity and brain activation will be measured while performing Task Switch.
Change in functional performance | At 5 years and at 3 months
  Between-group magnitude of change in sum time of all tasks in the Timed Instrumental Activities of Daily Living (TIADL). Higher scores indicate greater impairment in functional performance.
Change in Depressive Symptoms | At 5 years and at 3 months
  Between-group magnitude of change in sum score using the self-report measure, Center for Epidemiologic Studies Depression Scale (CES-D). The scoring range is 0-60. Higher scores indicate the presence of more symptomatology.
Blood-based Biomarker for Alzheimer's Disease | At 5 years
  Group differences in the P-tau181, Aβ1-42/Aβ1-40 concentrations

OTHER OUTCOMES:
Change in Stress | At 5 years and at 3 months
  Between-group magnitude of change in sum score using the self-report measure, Perceived Stress Scale (PSS-10). The scoring range is 0-40. Higher scores indicate higher perceived stress.
Change in Self-Efficacy | At 5 years and at 3 months
  Between-group magnitude of change in sum score using the self-report measure, Self-Efficacy Survey. The scoring range is 10-40. Lower scores indicate lower self efficacy.
Change in Life Satisfaction | At 5 years and at 3 months
  Between-group magnitude of change in sum score using the self-report measure, Life Satisfaction Scale. The scoring range is 5-35. Lower scores indicate lower life satisfaction.
Change in Physical Activity | At 5 years and at 3 months
  Change in total score based on weekly self-report dairy about physical activity during training period.
Change in Diet | At 5 years and at 3 months
  Change in total score based on weekly self-report dairy about diet during training period.
Change in Social Activity | At 5 years and at 3 months
  Change in total score based on weekly self-report dairy about social activity during training period.
Change in Sleep | At 5 years and at 3 months
  Change in total score based on weekly self-report dairy about sleep during training period.
Change in Functional Abilities | At 5 years and at 3 months
  Change in total score based on weekly self-report dairy about functional abilities during training period.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Kyu Lee, PhD, Principal Investigator — Posit Science Corporation
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - University of Texas at Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No